CLINICAL TRIAL: NCT06232954
Title: Evaluation of the Protective Efficacy of a Spatial Repellent to Reduce Malaria Prevalence in Children ≤ 5 Years of Age in Uganda: Study Protocol for a Cluster-randomized Double-blinded Control Trial: The Mossie-GO Trial
Brief Title: Evaluation of the Protective Efficacy of a Spatial Repellent to Reduce Malaria Prevalence in Uganda
Acronym: Mossie-GO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Power Limited (Industry)
Collaborators: Malaria Consortium (Other); ARCTECH INNOVATION LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1577
Record Dates: First submitted 2024-01-04; First posted 2024-01-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Malaria; Mosquito-Borne Disease
Keywords: malaria; spatial repellent; vector control; transfluthrin; randomised control trial
MeSH Terms: conditions — Malaria; Mosquito-Borne Diseases

STUDY DESIGN:
Intervention Model Description: Cluster-randomised placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: In exception of the data management personnel responsible for coordinating the manufacture and distribution of the Mossie-GO and independent statistician preparing the Data Safety and Monitoring Board (DSMB) report, all study staff will remain blinded to the household treatment allocation, until the completion of data collection and the locking of the database at the end of the study. Unblinded study staff will have no role in study implementation or outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All recruited households within the intervention arm will receive the Mossie-Go device containing transfluthrin treated discs and will be provided with refill transfluthrin discs at monthly intervals to provide sustained protection.
  Interventions: Device: Mossie-Go containing treated transfluthrin disc
- Control (Placebo Comparator): All recruited households within the control arm will receive the Mossie-Go device containing untreated blank discs and will be provided with refill untreated blank discs at monthly intervals.
  Interventions: Device: Mossie-Go containing untreated blank disc

INTERVENTIONS:
Device: Mossie-Go containing treated transfluthrin disc — The Mossie-GO repellent device is approximately 8 cm3 and can be fitted with repellent discs impregnated with transfluthrin and a carrier oil. These discs sit above a fan that is powered by a small motor charged by solar energy. The device is expected to both prevent bites and cause some mortality to mosquitoes when switched on for 8-12 hours overnight for up to 1 calendar month. The discs then need to be replaced.
  Arms: Intervention
Device: Mossie-Go containing untreated blank disc — The Mossie-GO repellent device is approximately 8 cm3 and can be fitted with a blank untreated disc. These discs sit above a fan that is powered by a small motor charged by solar energy. The device containing the untreated disc is not expected to prevent mosquito bites. The discs will still be replaced monthly for blinding purposes.
  Arms: Control

SUMMARY:
A cluster-randomized double-blinded control trial will be conducted in Uganda to demonstrate and quantify the protective efficacy (PE) of Mossie-GO, an active spatial repellent system disseminating transfluthrin, in reducing the prevalence of malaria in children ≤ 5 years of age, as determined by RDT positivity and confirmed by microscopy. The study's secondary objective is to measure the diversionary impact of the intervention on locally unprotected individuals and impact of the intervention on entomological correlates of transmission including vector densities, host seeking behaviour and insecticide resistance. This will be conducted using Centre of Disease Control (CDC) light traps in households, human landing catches and World Health Organisation (WHO) tube tests. Further data collection include household behavioural surveys, air sampling to quantify concentration of transfluthrin present in air, acceptability surveys and intervention safety monitoring.

Recruited households will be monitored across baseline data collection and followed up for 2 disease transmission seasons, for up to 18 months. The devices will be distributed to all consented eligible households in the two study arms: intervention and control. Intervention arm devices will be provided with transfluthrin treated discs and refill transfluthrin discs at frequent enough intervals to provide sustained protection. Households in the control arm will receive blank discs with no active ingredient. Households will be asked to continue using other malaria prevention practices, such as the use of bed nets, as recommended by national policy.

DETAILED DESCRIPTION:
The impact of Mossie-GO on malaria cases will be determined through a blinded cluster randomized trial in malaria endemic settings. The device will be distributed to all consented eligible households in the two study arms: intervention and control. Intervention arm devices will be provided with transfluthrin treated discs and refill transfluthrin discs at frequent enough intervals to provide sustained protection. Households in the control arm will receive blank discs with no active ingredient and refill blank discs to maintain study blinding.

The Mossie-GO repellent device is approximately 8 cm3 and can be fitted with repellent discs impregnated with transfluthrin and a carrier oil. These discs sit above a fan that is powered by a small motor charged by solar energy. The device is expected to both prevent bites and cause some mortality to mosquitoes when switched on for 8-12 hours overnight for up to 1 calendar month. The discs then need to be replaced. One Mossie-GO device will be provided per household, along with a solar cell unit that will be connected to the Mossie-GO unit and must be placed in direct sunlight to charge the Mossie-Go unit during the day, for use in the evening. Households will be asked to continue using other malaria prevention practices, such as bed nets, as recommended by national policy.

At baseline, Mossie-GO will be distributed at the household level and should be placed in the room of the participant enrolled into the study (child ≤ 5 years of age) while they are sleeping. At the same time a baseline survey will be conducted and children ≤ 5 years of age will be tested for malaria using RDTs and microscopy, to determine baseline malaria prevalence. At this time, household surveys will also be conducted to classify housing structure and collect other variables which may impact the efficacy of the intervention. Following this period, sample size estimates may be adjusted based on malaria prevalence. All recruited households will be monitored at 6-monthly intervals and malaria testing will be done among children ≤ 5 years of age with RDTs and microscopy over a period of up to 18 months. Indoor light traps will be installed in selected households for approximately 3-4 nights in the 6 month intervals and run from 6pm to 7 am to collect mosquitoes indoors, and human landing catches will be conducted. Air sampling will also be conducted alongside mosquito collections to quantify the concentrations of transfluthrin in the air and to help inform entomological and epidemiological outcomes. An acceptability survey will also be conducted at the final data collection time point

The unit of randomization is a cluster, which is defined as a discrete village or area containing a minimum of 100 households. Clusters will be divided into core and buffer zones. Twenty eight clusters will be identified per study arm (treatment and control), thus fifty six clusters will be selected in total. Households within the core zone of clusters will receive the Mossie-GO device (intervention or control). Households within the buffer zones will not receive the Mossie-GO. While all households within the core zone of the cluster are receiving the device, they will not all be sampled for the evaluation of the primary objective (PE). Only a total of 100 eligible, consenting households will be sampled within the core zones. Household surveys will also be conducted in these 100 households. For the evaluation of the secondary outcomes, a subset of houses will be selected. Diversionary impact: 100 households in buffer zone; entomological sampling: 10% of households in core zone; air sampling 1 household every 500m in core zone.

The primary outcome (PE) will be compared between arms using logistic regression with a random effect for study cluster and adverse event data will be collected and summarised.

ELIGIBILITY:
Inclusion Criteria:

Cluster level:

Number of households > 100

Household level:

Presence of a child ≤ 5 years of age at point of enrolment in the study

Adult head of household agrees to receiving and using the device as per manual instructions

Adult head of household agrees to data collection visits and household surveys

Children within household sleeps in cluster > 90% of nights during any given month

Individual level:

≤ 5 years of age when enrolled into the study

No plans for extended travel (> 1 month) outside of home during study

Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial

Provision of informed consent form (ICF) by the parent(s) or guardian

Participants not on regular malaria prophylaxis

Exclusion Criteria:

Cluster level:

Number of households < 100

Household level:

Presence of a child > 5 years of age at point of enrolment in the study

Adult head of household does not agree to data collection visits and household surveys

Children within household sleeps in cluster < 90% of nights during any given month

Households where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).

Individual level:

>5 years of age when enrolled into the study

Plans for extended travel (> 1 month) outside of home during study

Participating or planned participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial

No provision of ICF signed by the parent(s) or guardian

Participants on regular malaria prophylaxis

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5600 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Malaria prevalence | 18 months
  Malaria prevalence among children ≤ 5 years of age as determined by Rapid Diagnostic Test (RDT) positivity and confirmed by microscopy.

SECONDARY OUTCOMES:
Assessment of the diversionary effect of spatial repellent in the buffer zone using RDT and microscopy | 18 months
  Clusters are defined as discrete villages with a core and buffer zone. Buffer zones will be approximately 2km from the outer perimeter of the core zone and will not receive the intervention. This buffer zone will mitigate against the diversionary impact in the instance where villages are split into multiple clusters. The diversionary impact of the intervention on mosquitoes to locally unprotected individuals will be evaluated by measuring the malaria prevalence among children ≤ 5 years of age as determined by Rapid Diagnostic Test (RDT) positivity and confirmed by microscopy in a subset of households in the buffer zones. Mosquito population density and human biting rate will also be measured in the buffer zones.
Entomological correlates of transmission | 18 months
  Mosquito species composition and population density in mosquitoes caught using indoor CDC-light traps and Anopheline-human contact (indoor and outdoor) using human biting rate (HBR) as an indicator for all anophelines. Measured by human-landing catch (HLC).
Household surveys | 18 months
  Household surveys to collect information on subject behaviour related to exposure to malaria and use of existing control tools
Air sampling | 18 months
  Quantification of the temporal changes in concentration of transfluthrin present in the air over the duration of its use and the impact of indoor temperature on the concentration
Safety of intervention | 18 months
  Safety of intervention through monitoring of adverse events (AEs) and serious adverse events (SAEs)
Acceptability survey | 18 months
  Acceptability of Mossie-GO in these communities

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, PhD, Principal Investigator — Arctech Innovation; Jane Achan, PhD, Principal Investigator — Malaria Consortium
Locations (1):
- Malaria Consortium, Jinja, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dennehy J, Dyall W, Jenkins A, Bradley J, Sserwanga A, Kigozi R, Bwanika JB, Nuwa A, Mawejje H, Turner MA, Wallace R, Lyle FGA, Hiscox A, Livesey AK, Logan JG, Achan J, Jones RT. Evaluation of the protective efficacy of a transfluthrin-based spatial repellent product to reduce malaria prevalence in Uganda: study protocol for a cluster-randomised double-blinded control trial-the Mossie-GO trial. Trials. 2026 Feb 3. doi: 10.1186/s13063-025-09365-w. Online ahead of print. PMID 41634736